CLINICAL TRIAL: NCT00343252
Title: The Effect of Teriparatide Compared With Risedronate on Back Pain in Postmenopausal Women With Osteoporotic Vertebral Fractures
Brief Title: Effect of Teriparatide Compared to Risedronate on Back Pain in Women With a Spine Fracture Caused by Osteoporosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 9041; B3D-MC-GHCY (Other: Eli Lilly and Company)
Record Dates: First submitted 2006-06-20; First posted 2006-06-22 (Estimated); Results first posted 2010-07-12 (Estimated); Last update posted 2011-05-26 (Estimated); Status verified 2011-05

CONDITIONS: Osteoporosis, Postmenopausal; Back Pain; Spinal Fracture
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Back Pain; Spinal Fractures | interventions — Teriparatide; Risedronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Teriparatide (Experimental): Teriparatide 20 micrograms (ug)/day, subcutaneous, 18 months plus once weekly oral placebo
  Interventions: Drug: teriparatide; Drug: placebo
- Risedronate (Active Comparator): Risedronate 35 milligrams (mg)/once weekly, oral, 18 months plus daily subcutaneous injection placebo
  Interventions: Drug: risedronate; Drug: placebo

INTERVENTIONS:
Drug: teriparatide — 20 ug/day, subcutaneous, 18 months
  Other Names: LY333334; Forteo; Forsteo
  Arms: Teriparatide
Drug: risedronate — 35 mg/once weekly, oral, 18 months
  Other Names: Actonel
  Arms: Risedronate
Drug: placebo — once weekly, oral, 18 months
  Other Names: LY333334; Forteo; Forsteo
  Arms: Teriparatide
Drug: placebo — daily, subcutaneous, 18 months
  Other Names: Actonel
  Arms: Risedronate

SUMMARY:
The purpose of the study is to determine if daily teriparatide reduces back pain more effectively than weekly risedronate in women with osteoporosis who have chronic back pain due to a spinal bone fracture.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women 45 years or older. No period for at least two years.
* History of back pain that started at least 2 months prior to the initial visit (likely due to spinal bone fracture determined by investigator).
* Minimum of one moderate spinal bone fracture.
* Beginning pain level of at least four on an eleven point scale.
* Bone Mineral Density (BMD) must meet criteria
* Able to read, understand, and administer self-questionnaires.
* Be willing and able to use a pen-injector to deliver the medication.

Exclusion Criteria:

* Are at increased risk for osteosarcoma.
* Have an active or suspected diseases that affects bone metabolism other than osteoporosis.
* Participants that already know that they will require procedures to repair their spinal bone fractures.
* Abnormal values of certain lab tests.
* Anything that would make it difficult to determine if the back pain was due to the fracture.
* Poor medical or psychiatric condition.
* Alcohol or drug abuse within a year of the study start.
* Certain malignant neoplasms in the 5 years prior to enrollment.
* Active liver disease or clinical jaundice.
* Significantly impaired renal function.
* History of nephrolithiasis or urolithiasis within 2 years prior to enrollment.
* Known contraindication or intolerance to risedronate and/or teriparatide therapy.
* Treatment with oral strontium or certain therapeutic doses of fluoride.

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 712 (Actual)
Dates: Start 2006-06; Primary Completion 2009-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT -5 hours, EST), Study Director — Eli Lilly and Company
Locations (72):
- United States (20):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Birmingham, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montgomery, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Peoria, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Laguna Hills, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oakland, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Farmington, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palm Harbor, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Decatur, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gainesville, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Morton Grove, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Urbandale, Iowa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Omaha, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cleveland, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seattle, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spokane, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beckley, West Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madison, Wisconsin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marshfield, Wisconsin
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires, Argentina
- Australia (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kogarah, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Randwick, Sydney, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Maroochydore, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Keswick, South Australia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Malvern East
- Belgium (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brussels
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ghent
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gozée
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leuven
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Liège
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tienen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yvoir
- Brazil (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Campinas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rio de Janeiro
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., São Paulo
- Canada (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vancouver, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winnipeg, Manitoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamilton, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montreal, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sainte-Foy, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Trois-Rivières, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saskatoon, Saskatchewan
- France (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Amiens
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orléans
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poitiers
- Germany (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Braunfels
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Frankfurt
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heidelberg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heinsberg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leipzig
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., München
- Italy (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Siena
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Treviglio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valeggio sul Mincio
- Mexico (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., León
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
- Puerto Rico (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ponce
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan
- Spain (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Granada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salamanca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valencia
- Sweden (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Malmo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Solna
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Umeå
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Uppsala

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 712 participants were randomized: 361 to teriparatide; 351 to risedronate. 2 participants did not receive drug. Only randomized participants who received at least 1 dose of drug were analyzed. At 18 months, reason for discontinuation was corrected from sponsor decision to entry criteria not met (1) and protocol violation (1) for 2 participants.
Period: All Randomized Participants
Arm/Group | Teriparatide | Risedronate
Started | 361 | 351
Completed | 259 | 269
Not Completed | 102 | 82
Period: 6 Months (All Treated Participants)
Arm/Group | Teriparatide | Risedronate
Started | 360 (361 participants were randomized but 1 did not receive study drug and was not analyzed.) | 350 (351 participants were randomized but 1 did not receive study drug and was not analyzed.)
Completed | 304 | 306
Not Completed | 56 | 44
Not completed — Adverse Event | 17 | 11
Not completed — Death | 0 | 2
Not completed — Entry Criteria Not Met | 10 | 8
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lost to Follow-up | 0 | 4
Not completed — Physician Decision | 1 | 3
Not completed — Protocol Violation | 2 | 2
Not completed — Sponsor Decision | 7 | 4
Not completed — Withdrawal by Subject | 19 | 9
Period: 12 Months (All Treated Participants)
Arm/Group | Teriparatide | Risedronate
Started | 360 (361 participants were randomized but 1 did not receive study drug and was not analyzed.) | 350 (351 participants were randomized but 1 did not receive study drug and was not analyzed.)
Completed | 274 (Completed 12 Months.) | 281 (Completed 12 Months.)
Not Completed | 86 | 69
Not completed — Adverse Event | 22 | 20
Not completed — Death | 3 | 3
Not completed — Entry Criteria Not Met | 10 | 10
Not completed — Lack of Efficacy | 1 | 1
Not completed — Lost to Follow-up | 1 | 5
Not completed — Physician Decision | 4 | 5
Not completed — Protocol Violation | 3 | 2
Not completed — Sponsor Decision | 9 | 6
Not completed — Withdrawal by Subject | 33 | 17
Period: 18 Months (All Treated Participants)
Arm/Group | Teriparatide | Risedronate
Started | 360 | 350
Completed | 259 | 269
Not Completed | 101 | 81
Not completed — Adverse Event | 31 | 23
Not completed — Death | 4 | 5
Not completed — Entry Criteria Not Met | 11 | 10
Not completed — Lack of Efficacy | 1 | 1
Not completed — Lost to Follow-up | 3 | 7
Not completed — Physician Decision | 4 | 7
Not completed — Protocol Violation | 3 | 3
Not completed — Sponsor Decision | 8 | 5
Not completed — Withdrawal by Subject | 36 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Teriparatide | Risedronate | Total
Number analyzed (Participants) | 360 | 350 | 710
Age Continuous [Mean (Standard Deviation); unit: years] | 70.54 (8.80) | 71.55 (8.12) | 71.04 (8.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 360 | 350 | 710
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic | 67 | 61 | 128
  African Descent | 2 | 3 | 5
  Caucasian | 285 | 286 | 571
  East Asian | 3 | 0 | 3
  Native American | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 50 | 48 | 98
  Argentina | 38 | 42 | 80
  Australia | 30 | 30 | 60
  Belgium | 7 | 6 | 13
  Brazil | 30 | 30 | 60
  Canada | 54 | 55 | 109
  France | 13 | 10 | 23
  Italy | 22 | 20 | 42
  Mexico | 23 | 23 | 46
  Puerto Rico | 12 | 10 | 22
  Spain | 32 | 32 | 64
  Sweden | 13 | 10 | 23
  Germany | 36 | 34 | 70
Number of Vertebral Fractures [Number; unit: participants] — A minimum of at least one moderate osteoporotic vertebral fracture was radiologically detected and vertebral fracture status was documented. A moderate vertebral fracture was defined as at least a 25% decrease in anterior, central, or posterior vertebral height (T4 to L4) as compared to the average height of adjacent vertebrae. This measure categorizes the number of vertebral fractures for each participant.
  participants
    Unknown or No Vertebral Fractures | 37 | 35 | 72
    1 Vertebral Fracture | 126 | 104 | 230
    >=2 Vertebral Fractures | 197 | 211 | 408
Prior Osteoporosis Drug Use [Number; unit: participants] — Participants answered yes or no regarding use of osteoporosis drugs prior to this study.
  participants
    Yes | 267 | 258 | 525
    No | 93 | 92 | 185
Severity of Vertebral Fracture [Number; unit: participants] — An experienced radiologist graded all vertebrae by visual inspection from normal (grade 0) to severely deformed (grade 3).
  participants
    Zero or Mild Severity (Grade 0) | 50 | 46 | 96
    Moderate Severity (Grade 2) | 160 | 166 | 326
    Severe (Grade 3) | 142 | 131 | 273
    Unknown or Not Reported | 8 | 7 | 15
Spinal Deformity Index [Number; unit: units on a scale] — Spinal deformity index is the summation of the severity of the vertebral fracture(s).
  units on a scale
    0 | 29 | 28 | 57
    1 | 11 | 16 | 27
    2 | 76 | 67 | 143
    >=3 | 236 | 232 | 468
    Unknown or Not Reported | 8 | 7 | 15
24-Hour Average Back Pain Score [Mean (Standard Deviation); unit: units on a scale] — 24-hour average back pain severity scores recorded daily on an 11-point numeric rating scale, an ordinal scale ranging from 0 (no pain) to 10 (worst possible pain). The 11-point scale is used for assessment of average back pain in the preceding 24 hours and is evaluated daily in the week prior to each scheduled study visit. Responders are defined as participants with at least a 30% reduction in the severity of average back pain from baseline to the specified last observation carried forward (LOCF) endpoint.
  units on a scale | 5.34 (1.86) | 5.40 (1.85) | 5.37 (1.85)
24-Hour Worst Back Pain Score [Mean (Standard Deviation); unit: units on a scale] — 24-hour worst back pain severity scores recorded daily on an 11-point numeric rating scale, an ordinal scale ranging from 0 (no pain) to 10 (worst possible pain). The 11-point scale is used for assessment of worst back pain in the preceding 24 hours and is evaluated daily in the week prior to each scheduled study visit. Responders are defined as participants with at least a 30% reduction in the severity of worst back pain from baseline to the 6-month last observation carried forward (LOCF) endpoint.
  units on a scale | 6.80 (1.63) | 6.91 (1.54) | 6.85 (1.59)
Body Mass Index [Mean (Standard Deviation); unit: kilograms/meters squared] — Body mass index is an estimate of body fat based on body weight divided by height squared.
  kilograms/meters squared | 26.30 (5.01) | 26.36 (4.91) | 26.33 (4.96)
Duration of Back Pain [Mean (Standard Deviation); unit: days] | 550.33 (918.18) | 550.88 (750.47) | 550.58 (842.78)
Height [Mean (Standard Deviation); unit: centimeters] | 154.82 (7.41) | 153.62 (7.86) | 154.23 (7.66)
Quality of Life Questionnaire of the European Foundation for Osteoporosis (QUALEFFO) Score [Mean (Standard Deviation); unit: units on a scale] — QUALEFFO is an osteoporosis-specific health instrument developed specifically for participants with vertebral deformities used to evaluate the effect of back pain and treatment on quality of life. The QUALEFFO questionnaire includes 41 items in 5 domains: pain, physical function, social function, general health perception, and mental function. The total score is calculated according to the scoring algorithm developed by the International Osteoporosis Foundation. Total scores are reported from 0 to 100, with lower scores corresponding to better quality of life.
  units on a scale | 47.08 (14.61) | 46.98 (14.39) | 47.03 (14.49)
Roland-Morris Disability Questionnaire Score [Mean (Standard Deviation); unit: units on a scale] — Roland-Morris Disability Questionnaire (RMDQ-24) is completed by the participant and measures the degree of disability due to back pain. The questionnaire consists of 24 statements and the participant is instructed to put a mark next to each appropriate statement. The number of statements marked is added up by the clinician and a total score is given. The total score ranges from 0 (no disability) to 24 (severe disability).
  units on a scale | 11.88 (5.47) | 12.12 (5.40) | 12.00 (5.44)
Weight [Mean (Standard Deviation); unit: kilograms] | 63.02 (12.70) | 62.27 (12.58) | 62.65 (12.63)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Responding With at Least a 30% Reduction in 24-Hour Worst Back Pain Severity at the 6-Month Endpoint
Description: 24-hour worst back pain severity scores recorded daily on an 11-point numeric rating scale, an ordinal scale ranging from 0 (no pain) to 10 (worst possible pain). The 11-point scale is used for assessment of worst back pain in the preceding 24 hours and is evaluated daily in the week prior to each scheduled study visit. Responders are defined as participants with at least a 30% reduction in the severity of worst back pain from baseline to the 6-month last observation carried forward (LOCF) endpoint.
Time Frame: 6 Months
Population: Number of intent-to-treat (ITT) participants who were randomized and received at least one dose of the study drug. Endpoint was on a last observation carried forward (LOCF) basis. Participants with non-missing outcomes were analyzed.
Measure: Number; unit: participants
Arm/Group | Teriparatide | Risedronate
Number analyzed (Participants) | 348 | 336
participants
  Responder to Treatment | 206 | 193
  Non-Responder to Treatment | 142 | 143
Statistical Analysis 1: Comparison: Teriparatide vs Risedronate; Tested the null hypothesis that there is no statistically significant difference between treatment groups in the proportion of participants with at least a 30% reduction in the severity of worst back pain from baseline to the 6-month endpoint; Test type: Superiority or Other; p = 0.642, Chi-square — All comparisons were conducted using a 2-sided significance level of 0.05; No adjustments for multiplicity were performed

2. Secondary Outcome: Number of Participants Responding With at Least a 30% Reduction in 24-Hour Worst Back Pain Severity at the 12-Month Endpoint
Description: 24-hour worst back pain severity scores recorded daily on an 11-point numeric rating scale, an ordinal scale ranging from 0 (no pain) to 10 (worst possible pain). The 11-point scale is used for assessment of worst back pain in the preceding 24 hours and is evaluated daily in the week prior to each scheduled study visit. Responders are defined as participants with at least a 30% reduction in the severity of worst back pain from baseline to the 12-month last observation carried forward (LOCF) endpoint.
Time Frame: 12 Months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Teriparatide | Risedronate
Number analyzed (Participants) | 348 | 336
participants
  Responder to Treatment | 233 | 220
  Non-Responder to Treatment | 115 | 116
Statistical Analysis 1: Comparison: Teriparatide vs Risedronate; Tested the null hypothesis that there is no statistically significant difference between treatment groups in the proportion of participants with at least a 30% reduction in the severity of worst back pain from baseline at the 12-month endpoint; Test type: Superiority or Other; p = 0.683, Chi-square — All comparisons were conducted using a 2-sided significance level of 0.05; No adjustments for multiplicity were performed

3. Secondary Outcome: Number of Participants Responding With at Least a 30% Reduction in 24-Hour Average Back Pain Severity at the 6-Month Endpoint
Description: 24-hour average back pain severity scores recorded daily on an 11-point numeric rating scale, an ordinal scale ranging from 0 (no pain) to 10 (worst possible pain). The 11-point scale is used for assessment of average back pain in the preceding 24 hours and is evaluated daily in the week prior to each scheduled study visit. Responders are defined as participants with at least a 30% reduction in the severity of average back pain from baseline to the 6-month last observation carried forward (LOCF) endpoint.
Time Frame: 6 Months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Teriparatide | Risedronate
Number analyzed (Participants) | 347 | 336
participants
  Responder to Treatment | 221 | 211
  Non-Responder to Treatment | 126 | 125
Statistical Analysis 1: Comparison: Teriparatide vs Risedronate; Tested the null hypothesis that there is no statistically significant difference between treatment groups in the proportion of participants with at least a 30% reduction in the severity of average back pain from baseline to the 6-month endpoint; Test type: Superiority or Other; p = 0.809, Chi-square — All comparisons were conducted using a 2-sided significance level of 0.05; No adjustments for multiplicity were performed

4. Secondary Outcome: Number of Participants Responding With at Least a 30% Reduction in 24-Hour Average Back Pain Severity at the 12-Month Endpoint
Description: 24-hour average back pain severity scores recorded daily on an 11-point numeric rating scale, an ordinal scale ranging from 0 (no pain) to 10 (worst possible pain). The 11-point scale is used for assessment of average back pain in the preceding 24 hours and is evaluated daily in the week prior to each scheduled study visit. Responders are defined as participants with at least a 30% reduction in the severity of average back pain from baseline to the 12-month last observation carried forward (LOCF) endpoint.
Time Frame: 12 Months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Teriparatide | Risedronate
Number analyzed (Participants) | 347 | 336
participants
  Responder to Treatment | 246 | 238
  Non-Responder to Treatment | 101 | 98
Statistical Analysis 1: Comparison: Teriparatide vs Risedronate; Tested the null hypothesis that there is no statistically significant difference between treatment groups in the proportion of participants with at least a 30% reduction in the severity of average back pain from baseline to the 12-month endpoint; Test type: Superiority or Other; p = 0.986, Chi-square — All comparisons were conducted using a 2-sided significance level of 0.05; No adjustments for multiplicity were performed

5. Secondary Outcome: Number of Participants With Time to First Occurrence of at Least 30% Reduction in 24-Hour Worst Back Pain up to 6 Months
Description: Time to first occurrence of >= 30% pain reduction in worst back pain from baseline to 6 months. Worst back pain is assessed using an 11-point numeric rating scale, an ordinal scale ranging from 0 (no pain) to 10 (worst possible pain), to rate the worst back pain experienced in the preceding 24 hours and is evaluated daily in the week prior to each scheduled study visit. The results are reported as the number of participants reporting at least a 30% reduction in the severity of worst back pain up to time (t) in days.
Time Frame: Days 0, 30, 60, 90, 120, 150, 180, 210, 240, 270, and 300
Population: Number of intent-to-treat (ITT) participants who were randomized and received at least one dose of the study drug. Participants with non-missing outcomes were analyzed.
Measure: Number; unit: participants
Arm/Group | Teriparatide | Risedronate
Number analyzed (Participants) | 348 | 336
participants
  Day 0 | 0 | 0
  Day 30 | 26 | 22
  Day 60 | 70 | 74
  Day 90 | 110 | 111
  Day 120 | 151 | 145
  Day 150 | 175 | 164
  Day 180 | 195 | 181
  Day 210 | 206 | 192
  Day 240 | 206 | 193
  Day 270 | 206 | 193
  Day 300 | 206 | 193
Statistical Analysis 1: Comparison: Teriparatide vs Risedronate; Tested the null hypothesis that there is no statistically significant difference between treatment groups in the time to first occurrence of a >=30% reduction in worst back pain at the 6-month endpoint; Test type: Superiority or Other; p = 0.746, Log Rank — Comparison of the Kaplan-Meier survival curves between treatment groups was conducted using log-rank, significance level of 0.05; No adjustments for multiplicity were performed; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.85 to 1.26]

6. Secondary Outcome: Number of Participants With Time to First Occurrence of at Least 30% Reduction in 24-Hour Worst Back Pain up to 12 Months
Description: Time to first occurrence of >= 30% pain reduction in worst back pain from baseline to 12 months. Worst back pain is assessed using an 11-point numeric rating scale, an ordinal scale ranging from 0 (no pain) to 10 (worst possible pain), to rate the worst back pain experienced in the preceding 24 hours and is evaluated daily in the week prior to each scheduled study visit. The results are reported as the number of participants reporting at least a 30% reduction in the severity of worst back pain up to time (t) in days.
Time Frame: Days 0, 60, 120, 180, 240, 300, 360, 420, 480, 540, and 600
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Teriparatide | Risedronate
Number analyzed (Participants) | 348 | 336
participants
  Day 0 | 0 | 0
  Day 60 | 70 | 74
  Day 120 | 151 | 145
  Day 180 | 195 | 181
  Day 240 | 206 | 193
  Day 300 | 224 | 206
  Day 360 | 226 | 209
  Day 420 | 233 | 220
  Day 480 | 233 | 220
  Day 540 | 233 | 220
  Day 600 | 233 | 220
Statistical Analysis 1: Comparison: Teriparatide vs Risedronate; Tested the null hypothesis that there is no statistically significant difference between treatment groups in the time to first occurrence of a >=30% reduction in worst back pain at the 12-month endpoint; Test type: Superiority or Other; p = 0.719, Log Rank — [p-value comment as in outcome 5, analysis 1]; No adjustments for multiplicity were performed; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.86 to 1.25]

7. Secondary Outcome: Number of Participants With Time to First Occurrence of at Least a 30% Reduction in 24-Hour Average Back Pain up to 6 Months
Description: Time to first occurrence of >=30% pain reduction in average back pain from baseline to 6 months. Average back pain is assessed using an 11-point numeric rating scale, an ordinal scale ranging from 0 (no pain) to 10 (worst possible pain), to rate the average back pain experienced in the preceding 24 hours and is evaluated daily in the week prior to each scheduled study visit. The results are reported as the number of participants reporting at least a 30% reduction in the severity of average back pain up to time (t) in days.
Time Frame: Days 0, 30, 60, 90, 120, 150, 180, 210, 240, 270, and 300
Population: Number of intent-to-treat (ITT) participants who were randomized and received at least one dose of the study drug. Participants with non-missing outcomes were analyzed. The results are reported as the number of participants reporting at least a 30% reduction in the severity of back pain after time (t) in days.
Measure: Number; unit: participants
Arm/Group | Teriparatide | Risedronate
Number analyzed (Participants) | 347 | 336
participants
  Day 0 | 0 | 0
  Day 30 | 40 | 33
  Day 60 | 91 | 86
  Day 90 | 136 | 130
  Day 120 | 175 | 162
  Day 150 | 199 | 178
  Day 180 | 212 | 200
  Day 210 | 221 | 210
  Day 240 | 221 | 211
  Day 270 | 221 | 211
  Day 300 | 221 | 211
Statistical Analysis 1: Comparison: Teriparatide vs Risedronate; Tested the null hypothesis that there is no statistically significant difference between treatment groups in the time to first occurrence of a >=30% reduction for average back pain at the 6-month endpoint; Test type: Superiority or Other; p = 0.681, Log Rank — [p-value comment as in outcome 5, analysis 1]; No adjustments for multiplicity were performed; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.86 to 1.26]

8. Secondary Outcome: Number of Participants With Time to First Occurrence of at Least a 30% Reduction in 24-Hour Average Back Pain up to 12 Months
Description: Time to first occurrence of >= 30% pain reduction in average back pain from baseline to 12 months. Average back pain is assessed using an 11-point numeric rating scale, an ordinal scale ranging from 0 (no pain) to 10 (worst possible pain), to rate the average back pain experienced in the preceding 24 hours and is evaluated daily in the week prior to each scheduled study visit. The results are reported as the number of participants reporting at least a 30% reduction in the severity of average back pain up to time (t) in days.
Time Frame: Days 0, 60, 120, 180, 240, 300, 360, 420, 480, 540, and 600
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Teriparatide | Risedronate
Number analyzed (Participants) | 347 | 336
participants
  Day 0 | 0 | 0
  Day 60 | 91 | 86
  Day 120 | 175 | 162
  Day 180 | 212 | 200
  Day 240 | 221 | 211
  Day 300 | 234 | 220
  Day 360 | 238 | 226
  Day 420 | 246 | 238
  Day 480 | 246 | 238
  Day 540 | 246 | 238
  Day 600 | 246 | 238
Statistical Analysis 1: Comparison: Teriparatide vs Risedronate; Tested the null hypothesis that there is no statistically significant difference between treatment groups in the time to first occurrence of a >=30% reduction in average back pain at the 12-month endpoint; Test type: Superiority or Other; p = 0.789, Log Rank — [p-value comment as in outcome 5, analysis 1]; No adjustments for multiplicity were performed; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.86 to 1.23]

9. Secondary Outcome: Change From Baseline to 3-Month Endpoint in the Roland-Morris Disability Questionnaire.
Description: Roland-Morris Disability Questionnaire (RMDQ-24) is completed by the participant and measures the degree of disability due to back pain. The questionnaire consists of 24 statements and the participant is instructed to put a mark next to each appropriate statement. The number of statements marked are added up by the clinician and a total score is given. The total score ranges from 0 (no disability) to 24 (severe disability).
Time Frame: Baseline, 3 Months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Teriparatide | Risedronate
Number analyzed (Participants) | 334 | 311
units on a scale | -1.42 (0.45) | -1.41 (0.45)
Statistical Analysis 1: Comparison: Teriparatide vs Risedronate; Tested the null hypothesis that there is no statistically significant difference between the treatment groups in the proportion of participants with a reduction in disability at the 3-month endpoint; Test type: Superiority or Other; p = 0.968, ANCOVA — No adjustments for multiplicity were performed; The model includes terms for treatment, pooled site, baseline glucocorticoid usage status (yes/no), and baseline score

10. Secondary Outcome: Change From Baseline to 6-Month Endpoint in the Roland-Morris Disability Questionnaire.
Description: as for outcome 9
Time Frame: Baseline, 6 Months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Teriparatide | Risedronate
Number analyzed (Participants) | 341 | 319
units on a scale | -1.58 (0.48) | -1.77 (0.48)
Statistical Analysis 1: Comparison: Teriparatide vs Risedronate; Tested the null hypothesis that there is no statistically significant difference between treatment groups in the proportion of participants with a reduction in disability at the 6-month endpoint; Test type: Superiority or Other; p = 0.568, ANCOVA — No adjustments for multiplicity were performed; The model includes terms for treatment, pooled site, baseline glucocorticoid usage status (yes/no), and baseline score

11. Secondary Outcome: Change From Baseline to 12-Month Endpoint in the Roland-Morris Disability Questionnaire.
Description: as for outcome 9
Time Frame: Baseline, 12 Months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Teriparatide | Risedronate
Number analyzed (Participants) | 343 | 322
units on a scale | -2.09 (0.54) | -2.12 (0.53)
Statistical Analysis 1: Comparison: Teriparatide vs Risedronate; Tested the null hypothesis that there is no statistically significant difference between treatment groups in the proportion of participants with a reduction in disability at the 12-month endpoint; Test type: Superiority or Other; p = 0.932, ANCOVA — No adjustments for multiplicity were performed; The model includes terms for treatment, pooled site, baseline glucocorticoid usage status (yes/no), and baseline score

12. Secondary Outcome: Change From Baseline to 6-Month Endpoint, European Foundation for Osteoporosis Quality of Life Instrument (QUALEFFO)
Description: QUALEFFO is an osteoporosis-specific health instrument developed specifically for participants with vertebral deformities used to evaluate the effect of back pain and treatment on quality of life. The QUALEFFO questionnaire includes 41 items in 5 domains: pain, physical function, social function, general health perception, and mental function. The total score is calculated according to the scoring algorithm developed by the International Osteoporosis Foundation. Total scores are reported from 0 to 100, with lower scores corresponding to better quality of life.
Time Frame: Baseline, 6 Months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Teriparatide | Risedronate
Number analyzed (Participants) | 344 | 326
units on a scale | -2.80 (1.11) | -2.63 (1.10)
Statistical Analysis 1: Comparison: Teriparatide vs Risedronate; Tested the null hypothesis that there is no statistically significant difference between treatment groups in the proportion of participants with an improvement in quality of life at the 6-month endpoint; Test type: Superiority or Other; p = 0.814, ANCOVA — No adjustments for multiplicity were performed; The model includes terms for treatment, pooled site, baseline glucocorticoid usage status (yes/no), and baseline score

13. Secondary Outcome: Change From Baseline to 12-Month Endpoint, European Foundation for Osteoporosis Quality of Life Instrument (QUALEFFO)
Description: as for outcome 12
Time Frame: Baseline, 12 Months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Teriparatide | Risedronate
Number analyzed (Participants) | 344 | 327
units on a scale | -5.74 (1.23) | -5.27 (1.22)
Statistical Analysis 1: Comparison: Teriparatide vs Risedronate; Tested the null hypothesis that there is no statistically significant difference between treatment groups in the proportion of participants with an improvement in quality of life at the 12-month endpoint; Test type: Superiority or Other; p = 0.572, ANCOVA — No adjustments for multiplicity were performed; The model includes terms for treatment, pooled site, baseline glucocorticoid usage status (yes/no), and baseline score

14. Secondary Outcome: Number of Participants With Adverse Events (Safety) During 12 Months
Description: Safety was assessed via serious adverse events and all other non-serious adverse events and the data are located in the Reported Adverse Events Section.
Time Frame: Baseline through 12 Months
Population: Intent-to-treat (ITT). ITT participants are randomized participants who received at least one dose of teriparatide or risedronate.
Measure: Number; unit: participants
Arm/Group | Teriparatide | Risedronate
Number analyzed (Participants) | 360 | 350
participants
  Serious Adverse Events | 39 | 50
  Adverse Events | 269 | 266

15. Secondary Outcome: Number of Participants With Adverse Events (Safety) During 18 Months
Description: Safety is assessed via serious adverse events and all other non-serious adverse events and the data are located in the Reported Adverse Events Section.
Time Frame: Baseline through 18 Months
Population: as for outcome 14
Measure: Number; unit: participants
Arm/Group | Teriparatide | Risedronate
Number analyzed (Participants) | 360 | 350
participants
  Serious Adverse Events | 55 | 66
  Adverse Events | 277 | 273

16. Secondary Outcome: Number of Participants Responding With at Least a 30% Reduction in 24-Hour Worst Back Pain Severity at the 18-Month Endpoint
Description: 24-hour worst back pain severity scores recorded daily on an 11-point numeric rating scale, an ordinal scale ranging from 0 (no pain) to 10 (worst possible pain). The 11-point scale is used for assessment of worst back pain in the preceding 24 hours and is evaluated daily in the week prior to each scheduled study visit. Responders are defined as participants with at least a 30% reduction in the severity of worst back pain from baseline to the 18-month last observation carried forward (LOCF) endpoint.
Time Frame: 18 Months
Population: Intent-to-treat (ITT). Participants are participants who were randomized and received at least one dose of the study drug.
Measure: Number; unit: participants
Arm/Group | Teriparatide | Risedronate
Number analyzed (Participants) | 360 | 349
participants
  Responder | 248 | 234
  Non-Responder | 112 | 115
Statistical Analysis 1: Comparison: Teriparatide vs Risedronate; Test type: Superiority or Other; p = 0.600, Chi-squared — P-value is for responder versus non-responder

17. Secondary Outcome: Number of Participants Responding With at Least a 30% Reduction in 24-Hour Average Back Pain Severity at the 18-Month Endpoint
Description: 24-hour average back pain severity scores recorded daily on an 11-point numeric rating scale, an ordinal scale ranging from 0 (no pain) to 10 (worst possible pain). The 11-point scale is used for assessment of average back pain in the preceding 24 hours and is evaluated daily in the week prior to each scheduled study visit. Responders are defined as participants with at least a 30% reduction in the severity of average back pain from baseline to the 18-month last observation carried forward (LOCF) endpoint.
Time Frame: 18 Months
Population: Intent-to-treat (ITT). ITT participants were participants who randomized and received at least one dose of the study drug.
Measure: Number; unit: participants
Arm/Group | Teriparatide | Risedronate
Number analyzed (Participants) | 360 | 349
participants
  Responder | 260 | 242
  Non-responder | 100 | 107
Statistical Analysis 1: Comparison: Teriparatide vs Risedronate; Test type: Superiority or Other; p = 0.399, Chi-squared — P-value is for responder versus non-responder

18. Secondary Outcome: Number of Participants With Time to First Occurrence of at Least 30% Reduction in 24-Hour Worst Back Pain up to 18 Months
Description: Time to first occurrence of >= 30% pain reduction in worst back pain from baseline to 18 months. Worst back pain is assessed using an 11-point numeric rating scale, an ordinal scale ranging from 0 (no pain) to 10 (worst possible pain), to rate the worst back pain experienced in the preceding 24 hours and is evaluated daily in the week prior to each scheduled study visit. The results are reported as the number of participants reporting at least a 30% reduction in the severity of worst back pain up to time (t) in days.
Time Frame: Baseline through 18 Months
Population: Analysis includes number of randomized intent-to-treat (ITT) participants in each treatment group with non-missing time.
Measure: Number; unit: participants
Arm/Group | Teriparatide | Risedronate
Number analyzed (Participants) | 360 | 349
participants | 248 | 234
Statistical Analysis 1: Comparison: Teriparatide vs Risedronate; Test type: Superiority or Other; p = 0.453, Log Rank; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.89 to 1.28]

19. Secondary Outcome: Number of Participants With Time to First Occurrence of at Least a 30% Reduction in 24-Hour Average Back Pain up to 18 Months
Description: Time to first occurrence of >=30% pain reduction in average back pain from baseline to 18 months. Average back pain is assessed using an 11-point numeric rating scale, an ordinal scale ranging from 0 (no pain) to 10 (worst possible pain), to rate the average back pain experienced in the preceding 24 hours and is evaluated daily in the week prior to each scheduled study visit. The results are reported as the number of participants reporting at least a 30% reduction in the severity of average back pain up to time (t) in days.
Time Frame: Baseline through 18 Months
Population: Randomized intent-to-treat (ITT) participants in each treatment group with non-missing time.
Measure: Number; unit: participants
Arm/Group | Teriparatide | Risedronate
Number analyzed (Participants) | 360 | 349
participants | 260 | 242
Statistical Analysis 1: Comparison: Teriparatide vs Risedronate; Test type: Superiority or Other; p = 0.353, Log Rank; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.91 to 1.30]

20. Secondary Outcome: Change From Baseline to 18-Month Endpoint in the Roland-Morris Disability Questionnaire.
Description: Roland-Morris Disability Questionnaire (RMDQ-24) is completed by the participant and measures the degree of disability due to back pain. The questionnaire consists of 24 statements and the participant is instructed to put a mark next to each appropriate statement. The number of statements marked are added up by the clinician and a total score is given. The total score ranges from 0 (no disability) to 24 (severe disability). Pooled site, baseline glucocorticoid usage status (yes/no) and baseline score were controlled for.
Time Frame: Baseline, 18 Months
Population: Intent-to-treat (ITT). Participants who were randomized and received at least one dose of the study drug.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Teriparatide | Risedronate
Number analyzed (Participants) | 343 | 323
units on a scale | -3.21 (0.54) | -3.19 (0.53)
Statistical Analysis 1: Comparison: Teriparatide vs Risedronate; Test type: Superiority or Other; p = 0.943, ANCOVA

21. Secondary Outcome: Change From Baseline to 18-Month Endpoint in European Foundation for Osteoporosis Quality of Life Instrument (QUALEFFO)
Description: as for outcome 12
Time Frame: Baseline, 18 Months
Population: Intent-to-treat (ITT). Participants who were randomized and received at least one dose of the study drug.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Teriparatide | Risedronate
Number analyzed (Participants) | 344 | 327
units on a scale | -5.67 (1.27) | -5.17 (1.26)
Statistical Analysis 1: Comparison: Teriparatide vs Risedronate; Test type: Superiority or Other; p = 0.553, ANCOVA

ADVERSE EVENTS:
Time Frame: Baseline to 18 Months
Arm/Group | Teriparatide | Risedronate
Serious Adverse Events (participants affected / at risk) | 55/360 | 66/350
Other Adverse Events (participants affected / at risk) | 277/360 | 273/350
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teriparatide (N=360) | Risedronate (N=350)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 3 (4)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0)
Bundle branch block left (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 2 (2)
Ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Oscillopsia (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (3)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumoperitoneum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tongue disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Chest pain (General disorders) | 1 (1) | 3 (3)
Death (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Sudden death (General disorders) | 0 (0) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biliary dilatation (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 3 (3) | 0 (0)
Hepatic lesion (Hepatobiliary disorders) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Blister infected (Infections and infestations) | 1 (1) | 0 (0)
Bronchiectasis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 4 (4)
Helicobacter gastritis (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster disseminated (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis acute (Infections and infestations) | 1 (1) | 0 (0)
Pelvic abscess (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 1 (2)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 1 (1)
Vaginal abscess (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (3)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 5 (5) | 11 (11)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fractured coccyx (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (3)
Hip fracture (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 3 (4) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (2) | 3 (3)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (3)
Sternal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Scleroderma (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myelodysplastic syndrome transformation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 6 (7)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Embolic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Hyperreflexia (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 2 (2) | 0 (0)
Myoclonus (Nervous system disorders) | 2 (2) | 0 (0)
Nystagmus (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 2 (2) | 0 (0)
Oliguria (Renal and urinary disorders) | 1 (1) | 0 (0)
Ovarian mass (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Activities of daily living impaired (Social circumstances) | 0 (0) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Vertebroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive emergency (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Raynaud's phenomenon (Vascular disorders) | 1 (1) | 0 (0)
Temporal arteritis (Vascular disorders) | 0 (0) | 2 (2)
Vasospasm (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teriparatide (N=360) | Risedronate (N=350)
Diarrhoea (Gastrointestinal disorders) | 16 (19) | 22 (28)
Nausea (Gastrointestinal disorders) | 29 (37) | 30 (38)
Vomiting (Gastrointestinal disorders) | 9 (10) | 19 (22)
Bronchitis (Infections and infestations) | 22 (29) | 25 (27)
Influenza (Infections and infestations) | 29 (34) | 30 (37)
Nasopharyngitis (Infections and infestations) | 30 (35) | 25 (32)
Upper respiratory tract infection (Infections and infestations) | 18 (25) | 14 (17)
Urinary tract infection (Infections and infestations) | 23 (29) | 18 (20)
Fall (Injury, poisoning and procedural complications) | 33 (33) | 26 (35)
Arthralgia (Musculoskeletal and connective tissue disorders) | 36 (51) | 42 (51)
Back pain (Musculoskeletal and connective tissue disorders) | 18 (19) | 21 (22)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 32 (36) | 15 (19)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 20 (21) | 15 (18)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 25 (34) | 27 (32)
Dizziness (Nervous system disorders) | 21 (23) | 19 (21)
Headache (Nervous system disorders) | 34 (44) | 24 (25)
Hypertension (Vascular disorders) | 22 (22) | 21 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days